CLINICAL TRIAL: NCT01720706
Title: Thermal Ablation With a Loosely Wound Helical Coil for Radiofrequency Treatment of Large Renal and Hepatic Tumors in Patients Undergoing Partial or Total Nephrectomy or Heptectomy
Brief Title: Thermal Ablation in Larger Liver and Kidney Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFA
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Liver and Kidney Tumours
Keywords: Liver tumour; Kidney tumour; Hepatectomy; Nephrectomy; Metastatic Colon Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute (Experimental): The RFA Loosely wound thermal coil electrode will be inserted directly or percutaneously into the lesion, depending on the imaging modality (US or CT guidance) and deployed with same method as previously described in the 'delayed group'. Energy will be delivered using the single timed heating cycle. Treatment will be monitored with B mode US. Once the cycle is completed, the probe will be removed and the planned surgery will continue with partial or radical nephrectomy.
  Interventions: Device: RFA Loosely wound thermal coil
- Delayed (Experimental): Using an electrically insulated 12ga introducer with trocar is inserted percutaneously into the renal tumor. The needle tip will be placed 20mm from the center of the target. The trocar is removed and co-axially (i.e. within the introducer), a core biopsy of the lesion is performed with a 14-18 gauge needle. The radiofrequency applicator with a 14ga cannula containing the RFA Loosely wound thermal coil electrode is then optimally positioned and locked into the introducer. On approximately day 6-10, a partial or radical nephrectomy will be performed in the usual way.
  Interventions: Device: RFA Loosely wound thermal coil

INTERVENTIONS:
Device: RFA Loosely wound thermal coil — This new device uses radiofrequency energy to destroy kidney or liver tumours. It is called radiofrequency ablation.
  This type of energy is simply an alternating current that passes from a coil (electrode) into the tissue causing heating of the tissue in the vicinity of the electrode.
  Other Names: Devicedeveloped by the University Health Network

SUMMARY:
This is a clinical research study designed to determine the safety and efficacy of the application of a unique interstitial radio frequency thermal therapy for the treatment of large tumours in the kidney or liver. The novel device offers patients a more effective therapy than conventional RFA and for patients with large tumours fewer number of treatments and needle insertion sites. The clinical treatment volumes (or sites of focal tumours) will be determined by a combination of biopsy and contrast enhanced CT imaging.

The study will assess if novel device can produce lesions in the liver or kidney in a controlled and predictable manner and with sufficient size to effectively manage disease progression in the organ. The extent of lesion size at a delivered power setting and treatment time will be measured with post-treatment CT or MRI and biopsy as measures of tissue response

DETAILED DESCRIPTION:
Our group has developed a novel, interstitial induction coil device that has been designed to coagulate large tumours (≥3cm) through a single needle insertion using heat in the range 55-90 ◦C. [31]Our system consists of a helical coil that is loosely wound inside the tumour tissue or phantom and excited with radiofrequency energy at 27.12 MHz. The coil is constructed from Nitinol, a shape memory alloy, to permit percutaneous deployment of the device from a cannulating delivery needle into the tumor target. This novel monopolar device has the potential to treat larger tumours with larger ablation zones (6cm x 4cm) with shorter treatment time, in both ex vivo and in vivo settings. In our previous pig studies our group has not seen a decrease in ablation volume compared to the ex vivo studies. The intent of this research proposal is to determine the safety and efficacy of the application of a unique interstitial coil electrode RF thermal therapy device for ablating large human renal and hepatic tumors under US or CT guidance.

2. Hypothesis

Interstitial thermal therapy in the form of RF energy delivered percutaneously under US or CT guidance with our newly developed novel coil electrode is a safe and effective method to ablate large renal and hepatic tumors. This is an alternative to immediate surgery or to surveillance with possible delayed treatment.

3. Objectives

3.1 To use the novel RF device and technique in liver tumor as developed in the porcine model to patients with heptacellular carcinoma by:

3.1.1 Establishing that RF electrodes can be accurately and safely placed in the desired location.

3.1.2 Establish the safety of energy application with the RF coil device including assessing effect on surrounding liver tissue.

3.1.3 Verifying that large (>2cm) liver tumors are effectively ablated with RF energy.

3.2 To apply the novel RF device and technique in kidney tumor ablation as developed in the porcine model to patients with renal cell carcinoma by:

3.2.1 Establishing that RF electrodes can be accurately and safely placed in the desired location.

3.1.4 Establish the safety of energy application with the RF coil device including assessing effect on surrounding kidney tissue.

3.2.2 Verifying that large (RFA Loosely wound thermal coil2cm) kidney tumors are effectively ablated with RF energy.

4. Sample Size and Methods

4.1 RF ablation of renal tumor by:

4.1.1 Sample

Six patients with a large (large T1a and T1b N0 M0 RCC ,> 2 cm in diameter), solid renal mass who are undergoing partial or radical nephrectomy deemed suitable for additional RFA will be eligible.

The patients will be evenly split between two groups, namely the 'acute' and 'delayed'. With the acute group, the study can meet its study objectives while minimizing the number of procedures and evaluate the safety of the device with the patient in an OR suite. However, it is difficult to predict tumor viability accurately based on cellular effects of the RF treatment when the lesion is excised immediately after. The purpose of a delayed group examines the full extent of histological thermal changes which do not occur until 6-7 days after the treatment. This group will also validate the feasibility of the device within the intended clinical setting of an interventional CT suite.

Patients who might be considered eligible for standard RFA or with irreversible coagulation defects, urinary tract infection and/or morbid obesity will be excluded.

Only patients eligible for surgery for tumour resection will be enrolled. Patients will not be randomised. The first 3 patients will go into the acute group (immediate arm). The reason for this is to have a controlled setting should an incidence arise. The patient will already be prepared for surgery, which will provide a more controlled environment, should there be a patient safety issue.

4.1.2 Methods (Delayed Group)

The patient is admitted in the morning to the Medical Surgical Day Unit at the Toronto General Hospital. Initial nursing assessment includes the documentation of vital signs and allergies, and obtaining intravenous access. The patient is transported to the Department of Medical Imaging, where care is provided by the Interventional Radiology team consisting of a Radiologist, Radiology Nurse, and Radiology Technologist. Informed consent and satisfactory blood work results (platelet count, INR, and PTT) are confirmed. Pre-treatment CBC and creatinine will be measured and a urinalysis will be performed. Intravenous sedation is given (midazolam, fentanyl, meperidine, and/or dimenhydrinate) during the continuous monitoring of the patient, which includes pulse oximetry and blood pressure readings.

The appropriate area is aseptically prepared and draped, and the procedure is performed under real-time US and CT guidance. Local anesthesia (e.g. 10 ml of 1% lidocaine) is administered via a 25 gauge needle.

To ensure surrounding structures are protected from thermal injury, a "hydro-dissection technique" may be applied which acts as a "thermal blanket" around the kidney proven to be safe, effective, reproducible and inexpensive.

Using an electrically insulated 12ga introducer with trocar is inserted percutaneously into the renal tumor. The needle tip will be placed 20mm from the center of the target. The trocar is removed and co-axially (i.e. within the introducer), a core biopsy of the lesion is performed with a 14-18 gauge needle. The radiofrequency applicator with a 14ga cannula containing the loosely wound coil electrode is then optimally positioned and locked into the introducer. Applicator is rotated to line up target with coil trajectory. Coil 'introducer pliers' are used to deliver the coil into the tissue. Four dispersive electrodes (grounding pads) are adhered on the thighs of the patient. The applicator is connected to the generator and grounding pads. Energy will be applied in a single heating cycle for 4-10 minutes at a power rating set between 125-200W based on manual feedback and size of target. Development of the thermal lesion will be monitored with real time B mode US. At the end of the procedure the coil electrode is retracted with aid of the 'rectractor pliers' and then applicator with introducer is removed.

US or CT imaging is used during and immediately after RF to ensure accuracy of the thermal lesion created and to exclude complications. After completion of the procedure, the patient is transported to the Medical Surgical Day Unit for observation, recovery, and further pain control as required. Immediate post-treatment CBC and serum creatinine levels will be measured. Urinalysis will be performed. The patient is discharged home accompanied by a relative or a friend approximately 4 hours after completion of the RF procedure.

A follow-up contrast-enhanced spiral CT scan will be performed on approximately post-treatment day 6-10 (prior to the surgery) to assess possible complications and to measure the size of the lesion and degree of enhancement. In addition, CBC, serum creatinine and urinalysis will be performed.

On approximately day 6-10, a partial or radical nephrectomy will be performed in the usual way. In the cases of partial nephrectomy, it is assumed that clear margins will be grossly visible around the tumors to aid in the resection through normal tissue.

The specimen will be sent to pathology where thermal lesion sizes will be measured by gross inspection. Histo-pathology using standard H&E and NADH will establish the boundaries of the thermal lesion and detect any viable cells within this region. It will also establish the extent of coagulative necrosis in the normal surrounding kidney tissue. Further follow-up of the patient will continue as per standard protocol for RCC.

4.1.3 Methods (Acute Group)

In either the image guided therapy operating room (MPOR) or in the routine operating room at Toronto General Hospital the patient will be put under general anaesthesia.. A needle core biopsy will be taken from the lesion and sent to pathology for routine examination to ensure that an accurate diagnosis can be made if the subsequent thermal therapy alters the appearance of the tissue. A "hydro-dissection technique" is then applied to ensure surrounding structures are protected from thermal injury, which acts as a "thermal blanket" around the kidney.

The RF electrode will be inserted directly or percutaneously into the lesion, depending on the imaging modality (US or CT guidance) and deployed with same method as previously described in the 'delayed group'. Energy will be delivered using the single timed heating cycle. Treatment will be monitored with B mode US. Once the cycle is completed, the probe will be removed and the planned surgery will continue with partial or radical nephrectomy.

The specimen will be sent to pathology and processed as above.

For patients that have an ultrasound guided procedure, the RFA procedure will be done in the routine operating room in an open fashion, the kidney will be exposed surgically in the usual way in anticipation of the partial or radical nephrectomy. The kidney tumour will be located by gross inspection, palpation and with the aid of intraoperative US if required. In this case, the RFA probe will be inserted directly into the lesion. For those patients that have a CT guided procedure along with US, the procedure will be done in the MPOR and the RFA probe will be inserted percutaneously into the lesion, prior to opening and exposing the kidney. If the surgery is unable to be performed in the MPOR, the patient will transferred to a routine operating room, while under general anesthetic, to have their surgery. They will be accompanied by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a solid renal mass who are undergoing partial or radical nephrectomy
* subjects with a solid hepatic masses of heptacellular carcinoma or metastatic liver tumour booked for partial or radical hepatectomy

Exclusion Criteria:

* irreversible coagulation defects,
* hepatic infection,
* no extra hepatic malignant disease,
* venous invasion and/or
* morbid obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
RF electrodes can be accurately and safely placed in the desired location | up to 10 days prior to surgery and up to 24 hrs after surgery
  this will be assessed during the surgery and once the tumour is removed and examined

SECONDARY OUTCOMES:
The safety of energy application with the RF coil device including assessing effect on surrounding liver tissue | up to 10 days prior to surgery and up to 24 hrs after surgery
  This will be assessed during the surgery and once the tumour is removed and examined
Verifying that large (>2cm) liver tumors are effectively ablated with RF energy | up to 24hrs after surgery
  Once the tumour is removed, the ablation field can be fully examined.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jewett, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No